CLINICAL TRIAL: NCT02154828
Title: Clinical Evaluation of Integrative Practices Units Infant and Child Care for Unit Children With Typical or Atypical Autism (AUTISM)
Acronym: AUTISM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0029
Record Dates: First submitted 2014-04-15; First posted 2014-06-03 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Autism
Keywords: Children; aged; 3 to 6 years
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Integrative practices: Children included in this project are children 3 to 6 years with diagnosis F84.0 F84.1 according to CIM-10.
  these children must be supported in care units that meet the criteria defined integrative practices.
  Interventions: Behavioral: Integrative practices

INTERVENTIONS:
Behavioral: Integrative practices

SUMMARY:
The research project is part of the evaluation of the therapeutic approaches in mental health. Its framework infant and juvenile units that have developed "integrative devices," taking into account recent advances in knowledge and providing care, education and pedagogical approach. The evolution of autistic children receiving these integrative devices is studied to determine the validity of the devices mentioned. The methodology is based on case studies in a natural situation. Clinicians are committed to network among themselves and with researchers in a multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 to 6 years with diagnosis F84.0 and F84.1 according to ICD-10. The diagnosis should be made according to the criteria established by the recommendations on the diagnosis (FFP / HAS 2005).
* Children supported in care units that meet the criteria defined integrative practices.
* Children receiving a volume of hours of intervention between two and four half-days per week.
* Written parental consent collection.

Exclusion Criteria:

* Presence of co-morbidities such epilepsia, serious organ damage, somatic and sensory.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 3 to 6 years with a diagnosis F84.0 and F84.1 according to CIM-10, supported in care units that meet the criteria defined integrative practices.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Developmental evolution in the Psycho Educative-Profil 3 (PEP 3) scale between Month 0 and Month 12 | Month 12 (score : success or failure or emergence)
  The main objective is to evaluate scare practices in autism for children 3 to 6 years

SECONDARY OUTCOMES:
Global evolution of children by ECA-R scale | Month 12 (score 0 to 4)
Global evolution thanks to CARS scale | Month 12 (score between 15 and 60)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole GARRET-GLOANEC, PH, Principal Investigator — Nantes University Hospital
Locations (21):
- France (21):
  - CHI Robert Ballanger, Aulnay-sous-Bois
  - Daumezon hospital, Bouguenais
  - Brest University Hospital, Brest
  - Brive Hospital, Brivé
  - CH du Vinatier, Bron
  - Inercomunal Center, Créteil
  - Fondation Vallée, Gentilly
  - CH Gonesse, Gonesse
  - HDJ Les Marmousets, Haguenau
  - ARSEAA - Centre de guidance, Labège
  - CH Saint-Marie, Le Puy-en-Velay
  - Lille University Hospital, Lille
  - EPSM de l'agglomération Lilloise, Mons-en-Barœul
  - Nantes University Hospital, Nantes
  - Niort Hospital, Niort
  - HDJ La Pomme, Paris
  - Hôpitaux de St Maurice, Paris
  - Unité de soins précoces HJ René Diatkine ASM13, Paris
  - Saint-Nazaire Hospital, Saint-Nazaire
  - Centre Hospitalier CESAME, Sainte-Gemmes-sur-Loire
  - Rouvray Hospital, Sotteville-lès-Rouen

REFERENCES:
- [Derived] Bettencourt C, Garret-Gloanec N, Pellerin H, Pere M, Squillante M, Roos-Weil F, Ferrand L, Pernel AS, Apter G, Cohen D. Migration is associated with baseline severity and progress over time in autism spectrum disorder: Evidence from a French prospective longitudinal study. PLoS One. 2022 Oct 6;17(10):e0272693. doi: 10.1371/journal.pone.0272693. eCollection 2022. PMID 36201564